CLINICAL TRIAL: NCT06505382
Title: Effects of Ultrasound-Guided Percutaneous Neuromodulation of the Saphenous Nerve for Pain Management and Functionality in Patellofemoral Pain Syndrome Patients: A Single-Blind Randomized Controlled Trial
Brief Title: Effects of Percutaneous Neuromouldation of the Saphenous Nerve in Patients With Patellofemoral Pain
Acronym: PNMSNPFP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Castro Rodriguez, Physical Therapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Saphenous Nerve
Record Dates: First submitted 2024-06-14; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Patellofemoral Pain
Keywords: ultrasound-guided percutaneous neuromodulation; saphenous nerve; pain; functionality; femoropatellar pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNM group (Experimental): Participants in the experimental PNM group will receive ultrasound-guided percutaneous neuromodulation of the saphenous nerve in the painful leg.
  In this study, a neurostimulation device ITO ES-160 will be used, where parameters of 2 Hz, 250 μs, and 16 minutes of continuous current will be set, with an appropriate intensity for subjects to perceive nerve stimulation along the path of the nerve (from the needle insertion point to the anterior aspect and below the knee), always ensuring it remains tolerable for them. No motor response will be observed. The black clip of channel 1 will be attached to the needle, and a TENS patch will be attached to the red clip.
  The interventions will be conducted 3 times, with 1 week between the first two and a 2-week interval between the second intervention and the third. All measurements will be taken before and after the procedure.
  Interventions: Diagnostic Test: Ultrasound-guided percutaneous neuromodulation
- NON-PNM group (Placebo Comparator): Participants in the control NON-PNM group will receive saphenous nerve puncture in the injured leg with subsequent placement of the clamps but without activating the electrostimulation function.
  The needle will remain without current for 16 minutes. The interventions will be conducted 3 times, with 1 week between the first two and a 2-week interval between the second intervention and the third. All measurements will be taken before and after the procedure.
  Interventions: Diagnostic Test: Ultrasound-guided percutaneous neuromodulation

INTERVENTIONS:
Diagnostic Test: Ultrasound-guided percutaneous neuromodulation — Percutaneous ultrasound-guided neuromodulation of the saphenous nerve in subjects with patellofemoral pain to assess its positive effects on pain and functionality.

SUMMARY:
The knee is a common source of musculoskeletal pain, with patellofemoral pain (PFP) standing out due to its high prevalence. This pain, frequent in adolescents and athletes, significantly impacts the quality of life by hindering daily activities such as climbing stairs and sitting for extended periods. Percutaneous neuromodulation of the saphenous nerve (PNM) emerges as a promising therapeutic approach in physiotherapy to alleviate these symptoms.

A randomized controlled clinical trial is proposed in adults with PFP. Participants will be divided into two groups: one will receive PNM of the saphenous nerve, while the other will be a control group receiving puncture without electrical stimulation. Pain, extension strength, and knee range of motion will be evaluated before and after the intervention using the AKPS scale. Three sessions will be conducted with specific intervals, and a follow-up assessment will be performed three months later.

DETAILED DESCRIPTION:
Introduction: The knee is a common source of musculoskeletal pain, with patellofemoral pain (PFP) being one of the most prevalent. The incidence of PFP varies with age and activity level, but its impact on quality of life by causing pain and reduced functionality is significant. A high prevalence has been observed in adolescents and athletes, with symptoms interfering in daily activities such as climbing stairs, squatting, or sitting for prolonged periods. Percutaneous neuromodulation of the saphenous nerve emerges as a promising therapeutic approach to improve these patients' symptoms within the scope of physiotherapy.

Objectives: To determine the efficacy of a physiotherapy protocol based on ultrasound-guided percutaneous neuromodulation of the saphenous nerve on functional performance and pain in patients with PFP.

Materials and Methods: A randomized controlled clinical trial is proposed in adults with PFP symptoms. Volunteers will be divided into two groups: an intervention group and a control group. The experimental group will receive ultrasound-guided percutaneous neuromodulation (PNM) of the saphenous nerve, while the control group will only receive nerve puncture without electrical stimulation. The AKPS scale will be used to evaluate pain before and after the intervention, as well as knee extension strength and range of motion. Three sessions will be conducted with a one-week interval between the first two and a two-week interval between the second and third sessions. Finally, a follow-up assessment of all items without intervention will be conducted at three months

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Knee pain in the anterior aspect or around the patella for at least 1 month, exacerbated by activities such as squatting, stair climbing, or prolonged sitting.
* Patients experiencing difficulty participating in sports due to pain.

Exclusion Criteria:

* Previous surgical intervention on the painful knee.
* Previous diagnosed knee pathology.
* Recent trauma or acute injury to the knee that may have led to the development of pain.
* Antiplatelet or anticoagulant therapy.
* Bilateral symptoms.
* Pain attributed to hypersensitivity of any peripheral nerve of the lower limbs or a positive electromyographic test.
* Lumbar spine pathologies (herniated disc, protrusion, etc.).
* Use of medications such as opioids or those with knee pain as a side effect.
* Belonephobia or any condition where percutaneous needle insertion is contraindicated.
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patellofemoral Pain | Before and after the puncture in all interventions. Up to 4 months
  To quantify "pain intensity," the Visual Analog Scale (VAS) will be used, allowing the patient to subjectively express the intensity of their pain. It consists of a 10 cm line, where one end represents complete absence of pain and the other end represents the maximum possible intensity of pain. The patient is asked to mark on the line the point that reflects their pain level, and the measurement is recorded in millimeters. Within the "pain intensity" variable, a sub-variable will record the difference in pain intensity before and after the invasive physiotherapy intervention, expressed as a percentage of relief. This approach will allow observation of pain evolution across different sessions and evaluation of the immediate effects of Percutaneous Ultrasound-guided Neuromodulation.

SECONDARY OUTCOMES:
Knee functionality | Before the puncture in all interventions. Up to 4 months
  The Kujala Knee Pain Score (AKPS) will be primarily measured, consisting of 13 items related to specific symptoms and aggravating activities associated with patellofemoral pain (e.g., stairs, squatting, prolonged sitting, pain). Participants select a response for each item. All items are scored on a weighted basis and summed to give a score out of 100, where 0 represents maximum disability and 100 represents no disability.

OTHER OUTCOMES:
Strength of the knee | Before and after the puncture in all interventions. Up to 4 months
  The subject to be evaluated will be positioned at the edge of the examination table with 85º of hip flexion and 90º of knee flexion. A padded strap will be placed 5 cm proximal to the lateral malleolus, attached to the pressure dynamometer, which in turn will be connected to a rigid strap. This setup allows for the assessment of isometric quadriceps contraction strength. Participants will perform a warm-up consisting of five submaximal and maximal isometric knee extension contractions (50-100% effort). Subsequently, they will perform 3 maximal isometric contractions lasting 3 seconds each, with 1 minute of rest between contractions. Finally, the highest force contraction will be recorded for data analysis.
The range of motion of the knee | Before and after the puncture in all interventions. Up to 4 months
  The measurement will be conducted with the volunteer in prone position. The pelvis will be stabilized by the weight of the volunteer, and the femur will be stabilized by the evaluating physiotherapist. From this starting position, the physiotherapist will instruct the volunteer to actively perform knee extension in the sagittal plane and coronal axis.
  For measuring the extension movement, the physiotherapist will place the universal goniometer with its axis at the lateral epicondyle of the femur, the fixed arm parallel to the longitudinal axis of the femur, and the movable arm parallel to the longitudinal axis of the fibula, towards the lateral malleolus. The movement will begin to be measured from 90 degrees of knee flexion, instructing the subject to extend the heel away from the buttock until maximum extension is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Castro-Rodriguez, B.S, Principal Investigator — University of Alcala; Samuel Fernandez-Carnero, PhD, Principal Investigator — University of Alcala
Locations (1):
- Campus Cientifico-Tecnologico UAH.Colegio de León c/ Libreros, 21, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neal BS, Lack SD, Lankhorst NE, Raye A, Morrissey D, van Middelkoop M. Risk factors for patellofemoral pain: a systematic review and meta-analysis. Br J Sports Med. 2019 Mar;53(5):270-281. doi: 10.1136/bjsports-2017-098890. Epub 2018 Sep 21. PMID 30242107
- [Background] Dutton RA, Khadavi MJ, Fredericson M. Patellofemoral Pain. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):31-52. doi: 10.1016/j.pmr.2015.08.002. PMID 26616176
- [Background] Boling MC, Padua DA, Marshall SW, Guskiewicz K, Pyne S, Beutler A. A prospective investigation of biomechanical risk factors for patellofemoral pain syndrome: the Joint Undertaking to Monitor and Prevent ACL Injury (JUMP-ACL) cohort. Am J Sports Med. 2009 Nov;37(11):2108-16. doi: 10.1177/0363546509337934. Epub 2009 Sep 24. PMID 19797162
- [Background] Thomee R, Renstrom P, Karlsson J, Grimby G. Patellofemoral pain syndrome in young women. II. Muscle function in patients and healthy controls. Scand J Med Sci Sports. 1995 Aug;5(4):245-51. PMID 7552770
- [Background] Jensen R, Kvale A, Baerheim A. Is pain in patellofemoral pain syndrome neuropathic? Clin J Pain. 2008 Jun;24(5):384-94. doi: 10.1097/AJP.0b013e3181658170. PMID 18496302
- [Background] De-la-Cruz-Torres B, Abuin-Porras V, Navarro-Flores E, Calvo-Lobo C, Romero-Morales C. Ultrasound-Guided Percutaneous Neuromodulation in Patients with Chronic Lateral Epicondylalgia: A Pilot Randomized Clinical Trial. Int J Environ Res Public Health. 2021 May 3;18(9):4877. doi: 10.3390/ijerph18094877. PMID 34063673
- [Background] Arias-Buria JL, Cleland JA, El Bachiri YR, Plaza-Manzano G, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrical Nerve Stimulation of the Radial Nerve for a Patient With Lateral Elbow Pain: A Case Report With a 2-Year Follow-up. J Orthop Sports Phys Ther. 2019 May;49(5):347-354. doi: 10.2519/jospt.2019.8570. Epub 2019 Jan 18. PMID 30658050
- [Background] San-Emeterio-Iglesias R, Minaya-Munoz F, Romero-Morales C, De-la-Cruz-Torres B. Correct Sciatic Nerve Management to Apply Ultrasound-Guided Percutaneous Neuromodulation in Patients With Chronic Low Back Pain: A Pilot Study. Neuromodulation. 2021 Aug;24(6):1067-1074. doi: 10.1111/ner.13396. Epub 2021 Apr 20. PMID 33876885
- [Background] Beltra P, Ruiz-Del-Portal I, Ortega FJ, Valdesuso R, Delicado-Miralles M, Velasco E. Sensorimotor effects of plasticity-inducing percutaneous peripheral nerve stimulation protocols: a blinded, randomized clinical trial. Eur J Pain. 2022 May;26(5):1039-1055. doi: 10.1002/ejp.1928. Epub 2022 Mar 3. PMID 35191131
- [Background] Rossi M, DeCarolis G, Liberatoscioli G, Iemma D, Nosella P, Nardi LF. A Novel Mini-invasive Approach to the Treatment of Neuropathic Pain: The PENS Study. Pain Physician. 2016 Jan;19(1):E121-8. PMID 26752480